CLINICAL TRIAL: NCT05545774
Title: Characterization of Neuromuscular Involvement in Late Adolescent and Adult Cystinosis Patients
Brief Title: Neuromuscular Characterisation in Late Adolescent and Adult Cystinosis Patients
Acronym: Cystinose
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cystinosis Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220694; 2022-A01649-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-08-02; First posted 2022-09-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cystinosis
Keywords: cystinosis; neuromuscular disorder; respiratory function; swallowing disorder
MeSH Terms: conditions — Cystinosis; Neuromuscular Diseases; Respiratory Aspiration; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A biological sample will be taken to assess renal function (creatininemia and glomerular filtration rate according to MDRD formula), thyroid function status (thyrotropin, TSH), diabetes detection (glycemia and glycated heamoglobin, HbA1c) and cystine leukocyte level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to evaluate the change in motor function of patients with cystinosis.

The secondary objectives of the study:

* assessment of the respiratory function;
* assessment of the muscle function;
* assessment of swallowing disorders;
* assessment radiologically of the muscular efficiency;
* assessment of lean mass / fat mass ratio;
* assessment of sleeping disorders;
* annual assessment of evolution of above functions.

All patients will be examined by experienced neuromuscular specialist (Pr Pascal Laforêt) and pulmonologist specialized in neuromuscular disorders (Pr Hélène Prigent). All evaluations will be performed in Raymond-Poincaré hospital (Teaching hospital of Assistance Publique - Hopitaux de Paris (APHP) and University of Paris-Saclay) neuromuscular center, coordinated by Pr Pascal Laforêt.

DETAILED DESCRIPTION:
This is a monocentric study. The enrollment will be performed as routine care in the department of neurology - neuromuscular center of Raymond Poincaré hospital (APHP).

Patients with cystinosis will be consecutively invited to participate in the study until 20 patients are included. This will avoid selection bias if any. For eligible non included patients, a specific non-identifying registry will be set-up with a very restricted number of variables indicative of disease severity at baseline, allowing for a comparison of included and non-included patients.

Participating cystinosis patients will be proposed to attend a one-day hospitalization. Evaluations will be performed during stable state upon baseline and during a follow-up visit 12 months later.

The study expected duration is 30 months with 18 months for patients' inclusion and 12 month-follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 16 years;
* Genetically confirmed diagnosis of cystinosis;
* Presenting motor deficiency of at least one muscle;
* Covered by health insurance.

Exclusion Criteria:

* Patient refusal;
* Foreign patients under AME health schema;
* Patients under legal protection;
* Pregnancy or breast-feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female, age ≥ 16 years, with confirmed diagnosis of cystinosis and presenting at least one motor deficiency, are eligibles for this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Change in motor function | 12 months
  By the Motor Function Measure (MFM) quantitative scale to measure the functional capacities of motors (0-100%, higher scores mean better capacities).

SECONDARY OUTCOMES:
Change in motor strength | 12 months
  By Manual Muscle Testing (MMT). Higher scores mean better outcome.
Change in walking capacity | 12 months
  by the 6-minutes walking test. Higher scores mean better outcome.
Change in the time to stand test | 12 months
  by the time to stand test. Higher scores mean better outcome.
Change in the the Box and block test | 12 months
  by the Box and block test. Higher scores mean better outcome.
Change in the Nine hole peg test | 12 months
  by the Nine hole peg test. Higher scores mean better outcome.
Change in Perdue pegboard test | 12 months
  by Perdue pegboard test. Higher scores mean better outcome.
Change in Kapanji test | 12 months
  by Kapanji test. Higher scores mean better outcome.
Change in pinch strength | 12 months
  by myopinch test. Higher value mean better outcome.
Change in grip strength | 12 months
  by myogrip test. Higher value mean better outcome.
Change in vital capacity | 12 months
  By spirometry. Higher value mean better outcome.
Change in inspiratory muscles function | 12 months
  By inspiratory maximal pressure. Higher value mean better outcome.
Change in expiratory muscles function | 12 months
  By expiratory maximal pressure. Higher value mean better outcome.
Change in diaphragmatic performance | 12 months
  By transdiaphragmatic pressures measurements. Higher value mean better outcome.
Incidence of breathing disorders during sleep | 12 months
  Detection by a polysomnography associated to capnography.
Change in ratio of fat mass/lean mass | 12 months
  By osteodensitometry
Change in swallowing function - Sidney Swallow questionnaire | 12 months
  By the Sidney Swallow questionnaire. Higher scores mean better outcome.
Change in swallowing function - Salassa and McHorney scores | 12 months
  By the Salassa and McHorney scores. Higher scores mean better outcome.
Change in swallowing function - time of swallowing | 12 months
  By the time of swallowing 80 ml of water (normal = 3-4 sec). Higher values mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laforêt, MD, PhD, Principal Investigator — Neurology Department, Raymond Poincaré Hospital, APHP; Hélène Prigent, MD, PhD, Study Director — Physiology department, Raymond Poincaré Hospital, APHP; Aude Servais, MD, PhD, Study Chair — Department of Nephrology and Transplantation, Necker-Enfants Malades University Hospital, APHP
Locations (2):
- France (2):
  - Neurology Department, Raymond-Poincaré hospital, APHP, Garches
  - Department of Nephrology and Transplantation Centre de référence des Maladies Rénales Héréditaires de l'Enfant et de l'Adulte, Necker-Enfants Malades University Hospital, APHP, Paris